CLINICAL TRIAL: NCT00314405
Title: Identification of Sentinel Lymph Node (SLN) in Breast Cancer Care: Clinical and Economical Evaluation of a Double Method Using Isotope and Methylene Blue Dye Injection.
Brief Title: Identification of Sentinel Lymph Nodes With Methylene Blue and Isotope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3157
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Infiltrative Breast Cancer
Keywords: sentinel lymph node; SLN; probe; breast cancer; lymphoscintigraphy; methylene blue dye
MeSH Terms: conditions — Breast Neoplasms | interventions — Methylene Blue; Surgical Procedures, Operative

INTERVENTIONS:
Drug: Methylene blue (1%)
Drug: Rhenium sulfure
Procedure: Surgical procedure
Procedure: Anatomo-pathologic procedure

SUMMARY:
The aim of this study is to evaluate the performance of a double labelling method using isotope and methylene blue dye injection to localize precisely Sentinel Lymph Node (SLN) in a series of 100 patients with infiltrative breast cancer justifying SLN excision. Method and patients: SLN excision will be performed on 100 patients treated for infiltrative breast cancer. After preoperative methylene blue dye injection and lymphoscintigraphy, individual localization of the radioactive and stained nodes will be performed. After the surgery, SLN will be submitted to serial analysis and immunohistochemistry. A comparison of the two methods and an economical evaluation of the complete procedure will be performed.

ELIGIBILITY:
Inclusion Criteria:

* patients with infiltrative breast cancer (diagnosed pre-operatively by core biopsy)
* approval and informed consent

Exclusion Criteria:

* chemotherapy
* locoregional radiotherapy
* prevalent axillary lymph node

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Determination of an optimized protocol for SLN identification, with a double method using isotope and methylene blue dye injection.

SECONDARY OUTCOMES:
Comparison of the results of SLN serial sectioning, with H&E and IHC staining
Economical evaluation of SLN procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Bellocq, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Gynécologie-Obstétrique, Hôpital Civil, Strasbourg, France

REFERENCES:
- [Result] Mathelin C, Croce S, Brasse D, Gairard B, Gharbi M, Andriamisandratsoa N, Bekaert V, Francis Z, Guyonnet JL, Huss D, Salvador S, Schaeffer R, Grucker D, Marin C, Bellocq JP. Methylene blue dye, an accurate dye for sentinel lymph node identification in early breast cancer. Anticancer Res. 2009 Oct;29(10):4119-25. PMID 19846959